CLINICAL TRIAL: NCT01060020
Title: Acute Hemodynamic Effects of Sildenafil in Patients With Severe Aortic Stenosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Brian Lindman, MD, Assistant Professor of Medicine, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-1780
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Aortic Stenosis
Keywords: Aortic valve stenosis; Sildenafil; Phosphodiesterase inhibitors; Hypertension, Pulmonary
MeSH Terms: conditions — Aortic Valve Stenosis; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sildenafil 40mg or 80mg (Experimental): A single oral dose of Sildenafil (either 40mg or 80mg) will be administered to a participant after baseline hemodynamics are measured in the catheterization lab. Each dose will be equally distributed among those with preserved (≥50%) and reduced (<50%) EF.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Single oral dose of 40mg or 80mg of Sildenafil
  Other Names: Revatio; Viagra

SUMMARY:
Pulmonary hypertension is common in patients with aortic stenosis and is associated with worse operative and long-term outcomes. Sildenafil has been shown to reduce pulmonary artery pressure and improve exercise performance in patients with left-sided heart failure, but this has not been tested in patients with aortic stenosis. We hypothesize that Sildenafil will produce a clinically significant decrease in pulmonary artery pressure in patients with severe aortic stenosis. The dose of Sildenafil that produces a significant decrease in pulmonary artery pressure will be safe and well tolerated in patients with and without a depressed ejection fraction.

DETAILED DESCRIPTION:
Patients with severe aortic stenosis referred for a clinically ordered right and left heart catheterization will be eligible. Twenty subjects will be enrolled: 10 patients will receive 40mg and 10 patients will receive 80mg; each dose will be equally distributed among those with preserved (≥50%) and reduced (<50%) EF. Subjects will get a baseline echo prior to the heart catheterization. Baseline invasive hemodynamic measurements will be performed using a Swan Ganz catheter. A single oral dose of sildenafil will then be administered (40mg or 80mg), followed by invasive hemodynamic measurements at 30 and 60 minutes. Also at 60 minutes, limited echocardiographic images will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis (AVA < 1.0 cm2)
* Referred for a clinically ordered right and left heart catheterization
* 18 years of age and older
* Able and willing to comply with all requirements of the study

Exclusion Criteria:

* Nitrate use within 24 hours
* SBP < 110 mmHg or MAP < 75 mmHg
* Severe mitral regurgitation
* Severe aortic regurgitation
* Increased risk of priapism
* Retinal or optic nerve problems or unexplained visual disturbance
* Alpha antagonists or cytochrome P450 3A4 inhibitors use within 24 hours
* Current or recent (≤ 30 days) acute coronary syndrome
* O2 sat < 90% on room air
* Females that are pregnant or believe they may be pregnant
* Any condition which the PI determines will place the subject at increased risk or is likely to yield unreliable hemodynamic data
* Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian R. Lindman, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Lindman BR, Zajarias A, Madrazo JA, Shah J, Gage BF, Novak E, Johnson SN, Chakinala MM, Hohn TA, Saghir M, Mann DL. Effects of phosphodiesterase type 5 inhibition on systemic and pulmonary hemodynamics and ventricular function in patients with severe symptomatic aortic stenosis. Circulation. 2012 May 15;125(19):2353-62. doi: 10.1161/CIRCULATIONAHA.111.081125. Epub 2012 Mar 25. PMID 22447809

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants stratified according to ejection fraction and randomized to either Sildenafil 40mg and 80mg Groups were combined into a single Arm/Group for analysis as pre-specified in the study protocol.
Groups:
- Sildenafil 40mg or 80mg: A single oral dose of Sildenafil (either 40mg or 80mg) will be administered to a participant after baseline hemodynamics are measured in the catheterization lab.
  Sildenafil: Single oral dose of 40mg or 80mg of Sildenafil
Period: Overall Study
Arm/Group | Sildenafil 40mg or 80mg
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sildenafil 40mg or 80mg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 86 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Mean Pulmonary Artery Pressure in the Whole Cohort.
Time Frame: Baseline and 60 minutes after drug administered
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Sildenafil 40mg or 80mg
Number analyzed (Participants) | 20
percent change | -25 [-32 to -21]

2. Secondary Outcome: Percent Change in Pulmonary Vascular Resistance in the Whole Cohort.
Time Frame: Baseline and 60 minutes after drug administered
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Sildenafil 40mg or 80mg
Number analyzed (Participants) | 20
percent change | -29 [-49 to -13]

3. Secondary Outcome: Percent Change in Cardiac Index.
Description: Cardiac index is cardiac output divided by body surface area.
Time Frame: Baseline and 60 minutes after drug administered
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Sildenafil 40mg or 80mg
Number analyzed (Participants) | 20
percent change | 4 [-4 to 12]

4. Secondary Outcome: Load Independent Index of Diastolic Filling.
Description: Measurements of the load independent index of diastolic filling were made with the parameterized diastolic filling formalism as previously described and validated with the use of transmitral Doppler E waves recorded during different respiratory states (regular breathing and held expiration and inspiration).
Time Frame: Baseline and 60 minutes after drug administered
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Sildenafil 40mg or 80mg
Number analyzed (Participants) | 20
unitless
  Baseline | 1.02 (0.07)
  60 minutes | 1.03 (0.08)

5. Secondary Outcome: Global Longitudinal Strain
Description: Global longitudinal strain was measured at baseline and 60 minutes after drug administration.
Time Frame: Baseline and 60 minutes after drug administered
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Sildenafil 40mg or 80mg
Number analyzed (Participants) | 20
percent
  Baseline | -13.5 (4.3)
  60 minutes | -13.8 (3.9)

ADVERSE EVENTS:
Arm/Group | Sildenafil 40mg or 80mg
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil 40mg or 80mg (N=20)
Hypotension (Cardiac disorders) | 2
SVT (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil 40mg or 80mg (N=20)
hypertensive emergency (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes